CLINICAL TRIAL: NCT00611052
Title: "Adolescents Coping With Stress": Prevention of Adolescent Major Depression in School Health Care
Brief Title: Prevention of Adolescent Major Depression
Acronym: CWSA-Fin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unsuccessful recruitment, failed training of the group leaders leading into lack of study groups
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: University of Helsinki (Other); University of Eastern Finland (Other); Kuopio University Hospital (Other); City of Vantaa (Other Government); City of Kuopio (Other Government); City of Turku (Other Government)
Responsible Party: Principal Investigator, Linnea Karlsson, senior researcher, Finnish Institute for Health and Welfare
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KTL423-0
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Depressive Disorder
Keywords: Depressive Disorder; Depressive Disorder, Major; Mental Health; Prevention
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Group cognitive intervention (the Adolescent Coping with Stress)
  Interventions: Behavioral: the Adolescent Coping with Stress
- 2 (Active Comparator): Treatment as usual
  Interventions: Behavioral: Treatment as usual
- 3 (Active Comparator): Healthy controls, receive usual health education in school health care
  Interventions: Other: usual health education

INTERVENTIONS:
Behavioral: the Adolescent Coping with Stress — A group cognitive intervention, manualized and highly structured. Includes 8 sessions (á 1.5 hours) and a booster session 6 months after termination of the actual intervention. Groups leaders are specifically trained for this course.
  Arms: 1
Behavioral: Treatment as usual — The usual treatment received by the adolescent with mild to moderate self-reported depressive symptoms in school health care.
  Arms: 2
Other: usual health education — usual health education given by the school nurses, targeted for healthy controls with no depressive symptoms according to the self-report scale
  Arms: 3

SUMMARY:
The main purpose of this study is to assess the effect of a cognitive group intervention on prevention of major depression in 14-15-year-old adolescents. Moreover, the effect on other selected mental health parameters are investigated.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate level depressive symptoms (RBDI self-report scale)
* adequate knowledge of the Finnish language
* informed consent from the adolescent (all) and his/her parent (under 15 years)
* healthy controls comprise subjects with no depressive symptoms

Exclusion Criteria:

* ongoing major depression, dysthymia or bipolar disorder
* ongoing other severe psychiatric illness precluding group participation
* mental retardation

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2008-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Major depression (diagnostic interview) High level of depressive symptoms (self-report scale) | 3 months, 6 months, 12months, 24 months, 36 months

SECONDARY OUTCOMES:
Suicidality (diagnostic interview, self-report scale) | 3 months, 6 months, 12 months, 24 months, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Mauri J Marttunen, Professor, Study Director — National Institute for Health nd Welfare, Dept of Mental Health and Substance Abuse Services
Locations (3):
- Finland (3):
  - Kuopio University Hospital and Kuopio University, Kuopio
  - Turku Primary Health care and Adolescent Psychiatric clinic, Turku
  - Vantaa Primary Health Care, Vantaa